CLINICAL TRIAL: NCT02139592
Title: Brentuximab Vedotin (ADCETRIS) IV Infusion - Special Drug Use Surveillance (All-case Surveillance) "Relapsed or Refractory CD30+ Hodgkin's Lymphoma or Anaplastic Large Cell Lymphoma"
Brief Title: Brentuximab Vedotin (Recombinant) for IV Infusion - Special Drug Use Surveillance (All-case Surveillance) "Relapsed or Refractory CD30+ Hodgkin's Lymphoma or Anaplastic Large Cell Lymphoma"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 291-011; JapicCTI-142455 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-04-17; First posted 2014-05-15 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Relapsed or Refractory CD30+ Hodgkin's Lymphoma or Anaplastic Large Cell Lymphoma
Keywords: Pharmacological therapy
MeSH Terms: conditions — Recurrence; Lymphoma, Large-Cell, Anaplastic | interventions — Brentuximab Vedotin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- brentuximab vedotin (recombinant) Intravenous infusion: Intravenous infusion of 1.8 mg/kg (body weight) of brentuximab vedotin (recombinant) administered once every three weeks
  Interventions: Drug: Brentuximab vedotin (recombinant)

INTERVENTIONS:
Drug: Brentuximab vedotin (recombinant) — Brentuximab vedotin (recombinant) for IV infusion
  Other Names: ADCETRIS IV Infusion 50 mg

SUMMARY:
The purpose of this study is to evaluate the safety of brentuximab vedotin (recombinant) for intravenous (IV) infusion (ADCETRIS IV Infusion 50 mg) in patients with relapsed/refractory CD30+ Hodgkin's lymphoma or anaplastic large cell lymphoma in the routine clinical setting, as well as to collect efficacy information for reference.

DETAILED DESCRIPTION:
The present survey was designed to evaluate the safety of brentuximab vedotin (recombinant) for IV infusion (ADCETRIS IV Infusion 50 mg) in patients with relapsed/refractory CD30+ Hodgkin's lymphoma or anaplastic large cell lymphoma in the routine clinical setting.

The usual adult dosage is 1.8 mg/kg (body weight) of brentuximab vedotin (recombinant) infused intravenously once every three weeks. The dose should be adjusted depending on the participant's condition. See the "PRECAUTIONS" section of the package insert.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated with brentuximab vedotin IV Infusion

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Relapsed or refractory CD30+ Hodgkin's lymphoma or anaplastic large cell lymphoma
Sampling Method: Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2014-04-17 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Osaka, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 198 investigative sites in Japan, from 17 April 2014 to 30 June 2017. Registration period for patients was from 17 April 2014 to 30 September 2014.
Pre-assignment Details: Participants with a historical diagnosis of relapsed/refractory CD30+ Hodgkin's lymphoma (HL) or anaplastic large cell lymphoma (ALCL) were enrolled. Participants received interventions as part of routine medical care.
Groups:
- Brentuximab Vedotin Infusion: Intravenous infusion of 1.8 mg/kg (body weight) of brentuximab vedotin (recombinant) administered once every three weeks. Participants received interventions as part of routine medical care.
Period: Overall Study
Arm/Group | Brentuximab Vedotin Infusion
Started | 292
Completed | 284
Not Completed | 8
Not completed — Case Report Forms Uncollected | 8

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set; The safety analysis set was defined as all participants who had the safety data defined on the protocol.
Arm/Group | Brentuximab Vedotin Infusion
Number analyzed (Participants) | 284
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.7 (19.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 184
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Japan | 284
Duration of Diagnosis of Hodgkin's Lymphoma (HL) or Anaplastic Large Cell Lymphoma (ALCL) [Count of Participants; unit: Participants] — Mean duration between start of study and first time of diagnosis of HL or ALCL was reported.
  Participants
    < 1 Year | 75
    >= 1 Year and < 3 Years | 105
    >= 3 Years and < 5 Years | 47
    >= 5 Years | 55
    Unknown | 2
Diagnosis [Count of Participants; unit: Participants]
  HL | 182
  ALCL | 101
  Others | 1
Recurrent and Refractory or Primary [Count of Participants; unit: Participants]
  Recurrent and Refractory | 281
  Primary | 3
Number of participants with CD30 Positive [Count of Participants; unit: Participants] | 284
ALK Positive or Negative [Count of Participants; unit: Participants] — Population: This baseline characteristic was analyzed only in participants who had been diagnosed with ALCL.
  Participants
    number analyzed (Participants) | 101
    ALK-Positive | 15
    ALK-Negative | 77
    Unknown | 9
Staging of Lymphoma [Count of Participants; unit: Participants] — Lymphoma is classified with following stages. Stage 1; Lymphoma in only 1 group of lymph nodes. Stage 2; Lymphoma in 2 or more groups of lymph nodes. Stage 3; There are lymph nodes that contain lymphoma on both sides of the diaphragm. Stage 4; The most advanced stage of lymphoma and lymphoma cells have spread to at least 1 body organ outside the lymphatic system.
  Participants
    Stage 1 | 10
    Stage 2 | 63
    Stage 3 | 70
    Stage 4 | 140
    Unknown | 1
B Symptom [Count of Participants; unit: Participants] — B symptom means participants have 1 or more these symptoms as following; Unintentional weight loss (more than 10% in the 6 months before you were diagnosed), Night sweats, Fevers (temperatures above 38 Celsius degrees).
  Participants
    Had B symptom | 124
    Had No B symptom | 160
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Following are ECOG grades. 0: Fully active, perform all pre-disease activities without restriction. 1: Restricted in physically strenuous activity but ambulatory, carry out work of a light or sedentary nature. 2: Ambulatory, capable of selfcare, unable to carry out any work activities, up and about more than (>) 50% of waking hours. 3: Capable of limited selfcare, confined to bed or chair >50% of waking hours. 4: Completely disabled, not capable of any selfcare, totally confined to bed or chair.
  Participants
    0 | 114
    1 | 104
    2 | 32
    3 | 19
    4 | 15
Healthcare Category [Count of Participants; unit: Participants] — Participants were categorized as outpatient and inpatient.
  Participants
    Outpatient | 45
    Inpatient | 238
    Unknown | 1
Predisposition to Hypersensitivity [Count of Participants; unit: Participants] — The baseline characteristic was analyzed in participants who had a liability or tendency to suffer from hypersensitivity.
  Participants
    Had Predisposition to Hypersensitivity | 51
    Had No Predisposition to Hypersensitivity | 231
    Unknown | 2
Hepatitis C Virus (HCV) Antibody Positive or Negative [Count of Participants; unit: Participants]
  HCV Antibody-Positive | 6
  HCV Antibody- Negative | 274
  Unknown | 4
Hepatitis B Surface (HBs) Antigen Positive or Negative [Count of Participants; unit: Participants]
  HBs Antigen-Positive | 6
  HBs Antigen-Negative | 271
  Unknown | 7
HBs Antibody Positive or Negative [Count of Participants; unit: Participants]
  HBs Antibody-Positive | 41
  HBs Antibody- Negative | 208
  Unknown | 35
Hepatitis B Virus Deoxyribonucleic Acid (HBV DNA) Positive or Negative [Count of Participants; unit: Participants]
  HBV DNA-Positive | 4
  HBV DNA-Negative | 106
  Unknown | 174
Medical History of Lung Disorder [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above.
  Participants
    Had Medical History | 9
    Had No Medical History | 275
Medical Complications of Lung Disorder [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had Presence of Medical Complications | 20
    Had No Presence of Medical Complications | 264
Medical History of Malignant Tumor [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above.
  Participants
    Had Presence of Medical History | 33
    Had No Presence of Medical History | 251
Medical Complications of Malignant Tumor [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had Presence of Medical Complications | 5
    Had No Presence of Medical Complications | 279
Medical History (Other Than Lung Disorder or Malignant Tumor) [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above.
  Participants
    Had Presence of Medical History | 68
    Had No Presence of Medical History | 216
Medical Complications (Other Than Lung Disorder or Malignant Tumor) [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had Presence of Medical Complications | 182
    Had No Presence of Medical Complications | 102
Concomitant Hepatic Disorder [Count of Participants; unit: Participants]
  Had Concomitant Hepatic Disorder | 25
  Had No Concomitant Hepatic Disorder | 259
Concomitant Renal Disorder [Count of Participants; unit: Participants]
  Had Concomitant Renal Disorder | 20
  Had No Concomitant Renal Disorder | 264
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 58.158 (13.0751)
BMI [Mean (Standard Deviation); unit: kg/meter (m)^2] — Body Mass Index = weight (kg)/[height (m)^2]
  kg/meter (m)^2 | 22.00 (3.991)
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 130
  Current Smoker | 16
  Ex-Smoker | 84
  Unknown | 54
Drug Therapy before Start of Brentuximab Vedotin Administration [Count of Participants; unit: Participants]
  Had Drug Therapy | 279
  Had No Drug Therapy | 5
Number of Regimens before Start of Brentuximab Vedotin Administration [Mean (Standard Deviation); unit: Number of Regimens] — Population: Population Analysis Description: This baseline characteristic was analyzed only in participants who had drug therapy before start of Brentuximab Vedotin administration.
  Number of Regimens
    number analyzed (Participants) | 279
    (all) | 2.7 (1.57)
Time in Days from Last Month of Previous Drug Therapy Regimen to First Cycle of Brentuximab Vendotin [Mean (Standard Deviation); unit: Days] | 299.1 (564.04)
Radiotherapy before Start of Brentuximab Vedotin Administration [Count of Participants; unit: Participants]
  Had Radiotherapy | 105
  Had No Radiotherapy | 179
Time in Days from Last Month of Most Recent Radiotherapy to First Cycle of Brentuximab Vendotin [Mean (Standard Deviation); unit: Days] — Population: Population Analysis Description: This baseline characteristic was analyzed only in participants who had radiotherapy before start of Brentuximab Vedotin administration. The number analyzed is the number of participants with data available for analysis.
  Days
    number analyzed (Participants) | 94
    (all) | 703.4 (954.27)
Hematopoietic Stem Cell Transplantation before Start of Brentuximab Vedotin Administration [Count of Participants; unit: Participants]
  Had No Hematopoietic Stem Cell Transplantation | 219
  Had Autologous Transplantation | 43
  Had Allogeneic Transplantation | 9
  Had Autologous and Allogeneic Transplantation | 12
  Unknown | 1
Number of Participants Who Were Not Pregnant [Count of Participants; unit: Participants] — Population: This baseline characteristic was analyzed only in female participants.
  Participants
    number analyzed (Participants) | 100
    (all) | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had One or More Adverse Events (AE) and Serious Adverse Events (SAE)
Time Frame: Up to Week 48 or until discontinuation of treatment
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin Infusion
Number analyzed (Participants) | 284
Participants
  AE | 238
  SAE | 97

2. Secondary Outcome: Percentage of Participants Who Achieve or Maintain Any Best Response
Description: Best response is defined as the cumulative numbers of participants who achieve each level of best response including partial response (PR), complete response uncertain (CRu) (when no positron emission tomography [PET] data are available), and complete response (CR) after each cycle of treatment. Reported data are divided into 4 populations; Hodgkin's lymphoma (HL) participants with PET data, HL participants without PET data, anaplastic large cell lymphoma (ALCL) participants with PET data, and ALCL participants without PET data. PET is used in cancer diagnosis and treatment.
Time Frame: Up to Week 48 or until discontinuation of treatment
Population: Efficacy assessment population; The efficacy assessment population was defined as participants who met the requirement of this study and had efficacy data available for analysis. The number analyzed is the number of participants with data available for analysis in the given timeframe.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Brentuximab Vedotin Infusion
Number analyzed (Participants) | 241
Percentage of participants
  HL Participants with PET Data: number analyzed (Participants) | 77
  HL Participants with PET Data | 64.9 [53.22 to 75.47]
  HL Participants without PET Data: number analyzed (Participants) | 85
  HL Participants without PET Data | 36.5 [26.29 to 47.62]
  ALCL Participants with PET Data: number analyzed (Participants) | 37
  ALCL Participants with PET Data | 67.6 [50.21 to 81.99]
  ALCL Participants without PET Data: number analyzed (Participants) | 42
  ALCL Participants without PET Data | 57.1 [40.96 to 72.28]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the period from the start of therapy in standard medical care to the time when death (regardless of the cause of death) is confirmed. Reported data as OS was point estimates of 1 year survival rate for HL and ALCL participants.
Time Frame: Up to Week 48 or until discontinuation of treatment
Population: Efficacy assessment population; The efficacy assessment population was defined as participants who met the requirement of this study and had efficacy data available for analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Brentuximab Vedotin Infusion
Number analyzed (Participants) | 280
Percentage of participants
  HL Participants: number analyzed (Participants) | 179
  HL Participants | 82.7 [75.4 to 88.0]
  ALCL Participants: number analyzed (Participants) | 101
  ALCL Participants | 79.3 [68.4 to 86.7]

ADVERSE EVENTS:
Time Frame: Up to Week 48 or until discontinuation of treatment
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. For data of "Other Adverse Events", participants may be represented in more than 1 category.
Arm/Group | Brentuximab Vedotin Infusion
All-Cause Mortality (participants affected / at risk) | 51/284
Serious Adverse Events (participants affected / at risk) | 97/284
Other Adverse Events (participants affected / at risk) | 238/284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin Infusion (N=284)
Bacteraemia (Infections and infestations) | 1
Epstein-Barr virus infection (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 2
Meningitis aseptic (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 9
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 5
Systemic candida (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Pneumonia fungal (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Herpes zoster disseminated (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 3
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21
Peripheral T-cell lymphoma unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gingival cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaplastic large-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13
Anaemia (Blood and lymphatic system disorders) | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Bone marrow failure (Blood and lymphatic system disorders) | 1
Graft versus host disease (Immune system disorders) | 1
Acute graft versus host disease (Immune system disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Altered state of consciousness (Nervous system disorders) | 2
Cerebral haemorrhage (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 6
Clonic convulsion (Nervous system disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cardiomegaly (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 13
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Generalised erythema (Skin and subcutaneous tissue disorders) | 1
Renal disorder (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 2
Blood creatine phosphokinase increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 2
Transaminases increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Weight increased (Investigations) | 1
Brain herniation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin Infusion (N=284)
Lymphopenia (Blood and lymphatic system disorders) | 22
Neutropenia (Blood and lymphatic system disorders) | 153
Thrombocytopenia (Blood and lymphatic system disorders) | 17
Peripheral sensory neuropathy (Nervous system disorders) | 129
Rash (Skin and subcutaneous tissue disorders) | 15
Pyrexia (General disorders) | 15
Infusion related reaction (Injury, poisoning and procedural complications) | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT02139592/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT02139592/SAP_001.pdf